CLINICAL TRIAL: NCT01239160
Title: At Home Evaluation of Two Pneumatic Compression Devices in the Treatment of Lower Extremity Lymphoedema(ACE: At Home Compression Evaluation)
Brief Title: Two Pneumatic Compression Devices in the Treatment of Lower Extremity Lymphedema
Acronym: ACE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Futility and underpowering of endpoint data
Sponsor: Tactile Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Flexitouch 1010
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-10

CONDITIONS: Lymphedema
Keywords: lymphedema; pneumatic compression device; randomised clinical trial; volume reduction
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Advanced PCD (Experimental): The use of an advanced PCD device to reduce and maintain limb volume
  Interventions: Device: Flexitouch System
- Simple PCD (Active Comparator): The use of the Simple PCD is to reduce and maintain limb volume
  Interventions: Device: Hydroven FPR

INTERVENTIONS:
Device: Flexitouch System — A segmental, programmable, gradient pneumatic compression device. It consists of a controller and garment set. The garments are constructed of nylon and have 27-32 chambers, depending upon garment size. The pressure setting is variable between "normal" and "increased." The device is intended to be used for 60 minutes per day
  Arms: Advanced PCD
Device: Hydroven FPR — The FH is an intermittent sequential external pneumatic compression system. The garment contains 3 compression chambers. The pressure range of the compressor device is 30-100 mmHg. It is intended to be used for 60 minutes per day.
  Arms: Simple PCD

SUMMARY:
The treatment of lymphedema has been a major focus of attention for physicians and scientists for several decades. At this time, no successful techniques have been developed to prevent lymphedema, and therefore, a great deal of emphasis is placed on treatment modalities that can lessen the severity and impede the progression of this debilitating condition.

The treatment on offer usually consists of a maintenance phase using compression garments and an intensive treatment phase, which includes the use of skin care, compression bandaging, exercise and manual lymphatic drainage (MLD). The intensive phase is usually described as complex decongestive therapy (CDT). This is time consuming and requires high resource usage. Pneumatic compression devices (PCD) offer and alternative to MLD and can be used by the patient. There are a number of devices on the market that are categorized into 1. without calibrated gradient compression 2. With calibrated gradient compression.

This trial will compare two PCDs, a simple device without calibrated compression, and an advanced device with calibrated compression, in the reduction of swelling and maintenance of reduced limb volume in 262 patients with lower limb lymphoedema. The primary end point will be limb volume reduction over 12 weeks of treatment, with secondary outcome after 24 weeks.

DETAILED DESCRIPTION:
This is a Multicentre, prospective, single (assessor) blind randomised study. The primary objective of the study is to assess volume reduction in the treatment of lymphoedematous legs with an advanced PCD compared to a simple PCD in patients with lower limb lymphoedema. The main outcome is the percentage volume reduction of the affected limb at end of treatment compared to baseline.

Secondary objectives of the study are Assessment of safety Quality of life Health economic parameters

In total 262 patients with leg lymphoedema will be enrolled into the study. Patients eligible for the study are those who suffer from late stage II and stage III according to the International Society of Lymphology lymphoedema staging. Lymphoedematous legs can be of primary or secondary origin and uni or bilaterally affected. Medical history will be taken at baseline.

Patients will be taught how to use the device they have been randomised to. Visits will then take place at weeks 1,4,8,12 and 24 weeks. The device will be used for up to 60 minutes each day on the trial limb. At each visit sequential circumferences of the affected and unaffected limbs will be measured with a tape measure.

All adverse events will be documented. At beginning and end of study quality of life questionnaires and health economic information will be completed by the patients.

At the Derby site assessment of tissue quality will be made using ultrasound and moisture meter to assess tissue fluid.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be ≥ 18 years old or legal age in host country.
* Subjects must have a diagnosis of primary or secondary late Stage 2 or 3 unilateral or bilateral lower extremity lymphoedema.
* At time of initial evaluation, individuals must be at least 3 months post-surgery, chemotherapy and/or radiation treatment for cancer if applicable.
* If subjects were treated in a clinic setting for lymphoedema (Phase 1 treatment) they must be at least 3 months post completion of their acute care.

Exclusion Criteria:

* Diagnosis of active or recurrent cancer, or less than 3 months at the time of initial evaluation from the completion of chemotherapy, radiation therapy or primary surgery for the treatment of cancer.
* Diagnosis of acute infection. The source of the infection must be treated for 2 weeks prior to admittance into the study.
* Diagnosis of acute thrombophlebitis (in last 2 months)
* Diagnosis of peripheral arterial disease (PAD): PAD is defined as an Ankle Brachial Index (ABI), of 0.7 or lower.
* Diagnosis of pulmonary embolism or deep vein thrombosis within the previous 6 months
* Diagnosis of pulmonary edema
* Diagnosis of congestive heart failure (uncontrolled)
* Diagnosis of chronic kidney disease with a Glomerular Filtration Rate (GFR) of less than 30 mls per minute.
* Patients with poorly controlled asthma (i.e. those with severe persistent symptoms throughout the day, night time awakenings several times per week, use of a beta2 agonist inhaler several times per day and those whose normal activity is extremely limited).
* Pregnancy
* Any condition where increased venous and lymphatic return is undesirable
* Inability or unwillingness to participate in all aspects of study protocol and/or inability to provide informed consent
* Currently participating in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2010-11-02 (Actual); Primary Completion 2011-10-26 (Actual); Study Completion 2012-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine J Moffatt, RN PhD, Study Chair — Nottingham Trent University; Vaughan Keeley, MD, Study Director — Derby Hospitals NHS Trust; Margaret Sneddon, RGN, Principal Investigator — University of Glasgow; Peter J Franks, PhD, Principal Investigator — Tactile Medical
Locations (22):
- United States (10):
  - Hope Research Institute, Phoenix, Arizona
  - Northwestern University, Chicago, Illinois
  - Prairie Education & Research Cooperative, Springfield, Illinois
  - University of Missouri-Columbia,Ellis Fischel Cancer Center, Lymphedema Therapy Clinic, Columbia, Missouri
  - Stony Brook University Medical Center, Stony Brook, New York
  - Carolinas Rehabilitation, Charlotte, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Greenville Hospital Systems, Greenville, South Carolina
  - Fletcher Allen Health Care, Inc., University of Vermont, Colchester, Vermont
- Flinders Medical Center, Adelaide, Australia
- United Kingdom (11):
  - LOROS Hospice, Leicester, Leics
  - King's Mill Hospital, Mansfield, Nottinghamshire
  - University of Glasgow, Glasgow, Scotland
  - Abertawe Bro Morgannwg University, Swansea, West Glamorgan
  - Royal Derby Hospital, Derby
  - St Oswalds Hospice, Gosforth
  - Kendal Lymphology Centre, Kendal
  - Norfolk and Norwich University, Norwich
  - Queens Medical Center, Nottingham
  - Lymphoedema Clinic, Singleton Hospital, Swansea
  - St Giles Hospice, Whittington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Not Assigned: Consented, but did withdrawn prior to being randomized into one of the treatment groups.
Period: Overall Study
Arm/Group | Advanced PCD | Simple PCD | Treatment Not Assigned
Started (Of the 238 patients "started", 64 APCD and 66 SPCD had reached the 12 week visit milestone at the time of the outcome analysis reported below. Results presented include 130 subjects who had completed the 12 week follow up (or who withdrew within 12 weeks) prior to the 26Oct2011 dataset.) | 114 | 114 | 10
Completed | 89 | 95 | 0
Not Completed | 25 | 19 | 10
Not completed — Lost to Follow-up | 3 | 5 | 0
Not completed — Withdrawal by Subject | 17 | 6 | 2
Not completed — Physician Decision | 5 | 7 | 2
Not completed — Early Termination Due to Study Closure | 0 | 1 | 6

BASELINE CHARACTERISTICS:
Population: Results presented include 130 subjects who had completed the 12 week follow up (or who withdrew within 12 weeks) prior to the 26Oct2011 dataset.
Groups:
- Total: Total of all reporting groups
Arm/Group | Advanced PCD | Simple PCD | Total
Number analyzed (Participants) | 64 | 66 | 130
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 47 | 43 | 90
  ≥ 65 years | 17 | 23 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 52 | 99
  Male | 17 | 14 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 60 | 64 | 124
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 59 | 61 | 120
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25
  United Kingdom | 51 | 54 | 105
Etiology of Lymphedema [Count of Participants; unit: Participants]
  Primary | 34 | 34 | 68
  Secondary | 30 | 32 | 62
Severity of Lymphedema [Count of Participants; unit: Participants] — Late stage 2 is defined as prolonged swelling spontaneously irreversible, pitting becomes difficult to produce, presence of fibrosis, history of infection, the difference in circumference is between 4 and 6 cm (at a single point of measurement).
  Stage 3, considered worse than stage 2, is defined as presence of skin folds, severe tissue induration (fibrosis and sclerosis), skin changes (papillomas, hyperkeratosis, lymph cysts, fistulas), the difference in circumference is between greater than 6 cm (at a single point of measurement).
  Participants
    Late Stage II | 59 | 61 | 120
    Stage III | 5 | 5 | 10
Hosiery Used [Count of Participants; unit: Participants]
  Yes | 47 | 48 | 95
  No | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Limb Volume Change Between Baseline and 12 Weeks of Treatment - ml
Description: Limb volume in ml as assessed using the tape measure method of collecting circumferential leg measurements to insert into the truncated cone formula for limb volume calculation. A positive score indicates volume reduction between baseline and the noted follow-up, while a negative score indicates volume increase.
Time Frame: Baseline to 12 weeks was the primary outcome; other time points included for informational purposes.
Population: Of the 238 patients "started" in Participant Flow, 64 APCD and 66 SPCD had reached the 12 week visit milestone at the time of the outcome analysis. Results presented include 130 subjects who had completed the 12 week follow up (or who withdrew within 12 weeks) prior to the 26Oct2011 dataset. Data analyzed for subjects with measures assessed at the noted timepoint. Subjects who missed a visit or who did not complete the assessment at the visit were excluded.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Advanced PCD | Simple PCD
Number analyzed (Participants) | 64 | 66
ml
  Change Baseline to 1-Week: number analyzed (Participants) | 60 | 64
  Change Baseline to 1-Week | -11.1 (652.3) | 75.3 (678.0)
  Change Baseline to 4-Week: number analyzed (Participants) | 61 | 62
  Change Baseline to 4-Week | 7.4 (636.3) | 99.7 (691.3)
  Change Baseline to 8-Week: number analyzed (Participants) | 57 | 57
  Change Baseline to 8-Week | 77.7 (756.6) | 167.9 (760.7)
  Change Baseline to 12-Week: number analyzed (Participants) | 54 | 57
  Change Baseline to 12-Week | 102.1 (724.5) | 216.1 (919.3)

2. Primary Outcome: Limb Volume Change Baseline to 12 Weeks of Treatment - Percent
Description: Limb volume (percent change from baseline) as assessed using the tape measure method of collecting circumferential leg measurements to insert into the truncated cone formula for limb volume calculation. A positive score indicates volume reduction between baseline and the noted follow-up, while a negative score indicates volume increase.
Time Frame: Baseline to 12 weeks was the primary outcome; other time points included for informational purposes.
Population: Of the 238 patients "started" in Participant Flow, 64 APCD and 66 SPCD had reached the 12 week visit milestone at the time of the outcome analysis. Results presented include 130 subjects who had completed the 12 week follow up (or who withdrew within 12 weeks) prior to the 26Oct2011 dataset. Data analyzed for subjects with measures assessed at the noted timepoint. Subjects who missed visits or who did not complete the assessment at the visit were excluded.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Advanced PCD | Simple PCD
Number analyzed (Participants) | 64 | 66
percent change from baseline
  Change Baseline to 1-Week: number analyzed (Participants) | 60 | 64
  Change Baseline to 1-Week | -0.4 (6.2) | 0.9 (5.8)
  Change Baseline to 4-Week: number analyzed (Participants) | 61 | 62
  Change Baseline to 4-Week | -0.1 (6.3) | 0.9 (5.9)
  Change Baseline to 8-Week: number analyzed (Participants) | 57 | 57
  Change Baseline to 8-Week | 0.2 (7.4) | 1.6 (6.8)
  Change Baseline to 12-Week: number analyzed (Participants) | 54 | 57
  Change Baseline to 12-Week | 0.6 (6.4) | 2.2 (7.6)

3. Secondary Outcome: Adverse Events - Totals
Description: Adverse and serious adverse events will be recorded for patients for the duration of their participation in the trial
Time Frame: Up to 24 weeks of treatment
Population: Of the 238 patients "started" in Participant Flow, 64 APCD and 66 SPCD had reached the 12 week visit milestone at the time of the outcome analysis. Results presented include 130 subjects who had completed the 12 week follow up (or who withdrew within 12 weeks) prior to the 26Oct2011 dataset.
Measure: Number; unit: number of events
Arm/Group | Advanced PCD | Simple PCD
Number analyzed (Participants) | 64 | 66
number of events
  Total Serious Adverse Events (SAE) | 3 | 3
  Device-Related SAE | 2 | 0
  Procedure-Related SAE | 0 | 1
  Unrelated SAE | 1 | 2
  Total Non-Serious Adverse Events (NSAE) | 34 | 24
  Device-Related NSAE | 13 | 8
  Procedure-Related NSAE | 12 | 5
  Unrelated NSAE | 9 | 11

ADVERSE EVENTS:
Time Frame: Adverse events reported below were collected from Baseline through 24 week visit.
Description: Systematic assessment included investigator and study personnel asking subjects at each study visit if they had experienced any AEs since their previous visit. Results presented include 130 subjects who had completed the 12 week follow up (or who withdrew within 12 weeks) prior to the 26Oct2011 dataset.
Arm/Group | Advanced PCD | Simple PCD
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/66
Serious Adverse Events (participants affected / at risk) | 3/64 | 3/66
Other Adverse Events (participants affected / at risk) | 25/64 | 15/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Advanced PCD (N=64) | Simple PCD (N=66)
Edema (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Study leg became markedly swollen (no cellulitis).
Pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Extreme shooting pain followed by swelling and hardness of the leg.
Cancer (General disorders) | 0 (0) | 1 (1) — New diagnosis of lung cancer.
Fractured legs (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Fractured legs from motor vehicle accident.
Discoloration of toes (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Breathlessness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Breathlessness and dizziness.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Advanced PCD (N=64) | Simple PCD (N=66)
Worsened swelling/Edema (Blood and lymphatic system disorders) | 6 (6) | 4 (4)
Vomiting/Diarrhea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Pain/Itching (General disorders) | 9 (9) | 7 (7)
Cellulitis/Infection (Infections and infestations) | 6 (6) | 4 (5)

LIMITATIONS AND CAVEATS:
Early termination DSMB recommendation on 23Jan2012 due to underpowered endpoint in 26Oct2011 dataset. Results presented include 130 subjects who had completed the 12 week follow up (or who withdrew within 12 weeks) prior to the 26Oct2011 dataset.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less